CLINICAL TRIAL: NCT03481881
Title: Pharmacokinetics of Drugs Administered to Children Per Standard of Care
Brief Title: Pharmacokinetics of Drugs Administered to Children
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00042519
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pediatric ALL
Keywords: pharmacokinetics
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Standard of care drug — This study is collecting PK data on children prescribed the following drugs of interest per standard of care: dexmedetomidine, bosentan, furosemide, chlorothiazide, ethacrynic acid, bumetanide, hydromorphone, tacrolimus, ampicillin, gentamicin, caffeine, fentanyl, midazolam, foscarnet, hydroxychloroquine, and moxifloxacin.

SUMMARY:
This is a prospective study of children <21 years of age with the goal of characterizing the PK of drugs administered per standard of care as prescribed by the treating caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Children (< 21 years of age) who are receiving understudied drugs of interest per standard of care as prescribed by their treating caregiver

Exclusion Criteria:

* Failure to obtain consent/assent (as indicated)

Ages: 0 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (<21 years of age) receiving drugs per standard of care as prescribed by treating caregiver
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-08-14 (Actual); Primary Completion 2033-08-14 (Estimated); Study Completion 2033-08-14 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) | Data will be collected throughout the hospital or outpatient stay up to 90 days

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Data will be collected throughout the hospital or outpatient stay up to 90 days
Time to achieve maximum concentration (Tmax) | Data will be collected throughout the hospital or outpatient stay up to 90 days
Absorption rate constant (ka) | Data will be collected throughout the hospital or outpatient stay up to 90 days
Elimination rate constant (kel) | Data will be collected throughout the hospital or outpatient stay up to 90 days
Half-life (t1/2) | Data will be collected throughout the hospital or outpatient stay up to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No